CLINICAL TRIAL: NCT05353049
Title: A Bathing Intervention Based on Basale Stimulation® for People With Moderate to Severe Dementia
Brief Title: How to Bathe a Person With Dementia? A Bathing Intervention Based on Basale Stimulation® for People With Moderate to Severe Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Salamanca (Other)
Collaborators: National Reference Centre for Alzheimer's and Dementia Care (CREA), Spain (Unknown)
Responsible Party: Principal Investigator, Jaime Unzueta Arce, Assistant Professor of Psychology, University of Salamanca
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Basale Stimulation bathing
Record Dates: First submitted 2022-03-28; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Patient Engagement; Behavioral Symptoms
MeSH Terms: conditions — Patient Participation; Behavioral Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bathing technique based on Basale Stimulation (Experimental)
  Interventions: Behavioral: Bathing technique based on Basale Stimulation
- Traditional bathing technique (No Intervention)

INTERVENTIONS:
Behavioral: Bathing technique based on Basale Stimulation — The relaxing somatic modelling technique will be applied, framed within the concept of Basal Stimulation®. To do this, the user remains seated and the parts of the body that are not being washed at that moment are covered with a towel, favouring the preservation of the user's privacy. The user is lathered up with soft mittens previously moistened with lukewarm water and lathered up. This process shall be carried out starting from the shoulder in a proximal to distal direction on the upper limbs, lower limbs and trunk (taking into account the sagittal anatomical plane) and in a cephalic to caudal direction (taking into account the transverse anatomical plane).
  Subsequently, rinsing is carried out following the same guidelines as described above, using moistened soft mittens. Finally, intimate hygiene is performed with a disposable soapy sponge and the soap is rinsed off again with moistened soft terrycloth mittens. Throughout the whole process, the activity is explained to the user.
  Arms: Bathing technique based on Basale Stimulation

SUMMARY:
Brief summary Resisted behaviours that occur during showering of People with Dementia (PwD) cause greater discomfort for caregivers and may occur as a result of embarrassment and shame that the person with dementia may be experiencing or even due to a moment of confusion or anxiety.

Therefore, it is considered particularly relevant and necessary to provide information and strategies to caregivers of PwD in order to manage the behavioural alterations produced during the shower.

One of the strategies currently used in clinical practice to improve the relationship between caregivers and users is the implementation of the Basale stimulation® concept.

The stimuli applied from Basale Stimulation® are related to 3 basic areas of development: somatic, vestibular and vibrational. In relation to the development of the showers, they will be carried out from the application of relaxing somatic modelling connected to the somatic area.

The aim of this study is to analyse the efficacy of an intervention based on the relaxing somatic modelling technique, framed within the Basale Stimulation® concept, to reduce behavioural disturbances and increase the involvement of the person with moderate to severe dementia during assisted showering.

The main caregivers of the PwD, who meet the inclusion criteria will be contacted by sending a study information sheet and an informed consent form. All family members will receive a call to clarify the concepts explained and the study methodology to be carried out.

The grooming sessions of all users whose relatives have signed the informed consent form, will be videotaped and a trained technician will fill in the questionnaires for each session based on the analysis of the videos of each intervention.

Six intervention sessions will be carried out with each user. An alternating treatment design will be used, applying condition A or B randomly and then counterbalancing. Condition A corresponds to a traditional shower according to the long-term care bathing and grooming protocol and condition B corresponds to the use of relaxing somatic modelling within Basale Stimulation®.

The first result obtained will be an increase in the appearance and frequency of behaviours that increase the engagement of the PwD and a decrease in the appearance and frequency of disengagement behaviours during the shower activity in the Basale Stimulation® application sessions. This result will be measured with the Involvement Register (RIE) (García-Soler et al., 2014), adding the measure of frequency of involvement behaviours on a likert scale.

The second expected outcome will be the decrease in the occurrence, frequency and intensity of behavioural disturbances during the Basale Stimulation®-based intervention showers. This outcome will be measured with a questionnaire based on the Neuropsychiatric Inventory Questionnaire (NPI-Q)(Boada et al., 2002) and the Agitated Behavior in Dementia scale (ABID) (Logsdon et al., 1999), recording the number of times a disruptive behaviour appears, the frequency with which it appears during the shower, and the intensity of the behaviour on a Likert scale.

In addition, the user's functional status measured with the Barthel Index, his cognitive status measured with the Mini-Mental State Examination and his behaviour through the Agitation Inventory of the Elderly will be taken into account.

Intervention description The relaxing somatic modelling technique will be applied, framed within the concept of Basal Stimulation®. To do this, the user remains seated and the parts of the body that are not being washed at that moment are covered with a towel, favouring the preservation of the user's privacy. The user is lathered up with soft mittens previously moistened with lukewarm water and lathered up. This process shall be carried out starting from the shoulder in a proximal to distal direction on the upper limbs, lower limbs and trunk (taking into account the sagittal anatomical plane) and in a cephalic to caudal direction (taking into account the transverse anatomical plane).

Subsequently, rinsing is carried out following the same guidelines as described above, using moistened soft mittens. Finally, intimate hygiene is performed with a disposable soapy sponge and the soap is rinsed off again with moistened soft terrycloth mittens. Throughout the whole process, the activity is explained to the user.

ELIGIBILITY:
Inclusion Criteria:

* 55 years old or older
* Moderate or severe dementia (GDS 5 or higher)
* Long term care patients
* Dependent for bathing

Exclusion Criteria:

* Mild Cognitive Impairment or dementia with GDS 4 or lower.
* Need 2 or more people for assisted bathing
* Independence for showering

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of Engagement Behaviour assessed with the Involvement Register (RIE) | Through study completion, an average of 2 years
  Assessment of the frequency of engagement behaviour during bathing (1-5 likert scale: "1" meaning a lower frequency of engagement behavioural while "5" means a higher frequency of engagement behaviour during bathing).
  Higher scores (higher frequency of engagement behaviour) mean a better outcome.

SECONDARY OUTCOMES:
Presence and frequency of behavioural symptoms assessed with the a Behavioral questionnaire based on the Neuropsychiatric Inventory Questionnaire (NPI-Q) and the Agitated Behavior in Dementia scale (ABID) | Through study completion, an average of 2 years
  Evaluation of the presence and frequency of behavioural symptoms during bathing (1-5 likert scale: "1" meaning lower frequency of behavioural symptoms while "5" means a higher frequency of behavioural symptoms during bathing).
  Higher scores (higher frequency of behaviour symptoms) mean a worse outcome. The aim is is to reduce the frequency or eliminate behaviour symptoms.

OTHER OUTCOMES:
Intensity of behavioural symptoms assessed with the a Behavioral questionnaire based on the Neuropsychiatric Inventory Questionnaire (NPI-Q) and the Agitated Behavior in Dementia scale (ABID) | Through study completion, an average of 2 years
  Assessment of the intensity of behavioural symptoms presented during bathing (1-3 likert scale. 1: low intensity, 2: medium intensity, 3: high intensity of behavioural symptoms during bathing).
  Higher scores (higher intensity of behaviour symptoms) mean a worse outcome. If behavioural symptoms can not be eliminated, the aim is is to reduce intensity of those symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Salamanca, Salamanca, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No